CLINICAL TRIAL: NCT03313076
Title: Pilot, Double-blind, Randomized Controlled, Multi-center Study of the Effects of Fish Oil and Vitamin D in the Prevention of Chronic Pain Following Major Thermal Burn Injury
Brief Title: Vitamin D and n-3 Polyunsaturated Fatty Acids (PUFAs) to Prevent Chronic Pain Following Major Thermal Burn Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19 global pandemic, and study funding period ended 7/31/2020.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-1971
Record Dates: First submitted 2017-09-20; First posted 2017-10-18 (Actual); Results first posted 2021-07-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2021-03

CONDITIONS: Chronic Pain Following Thermal Burn Injury
Keywords: burn injury; thermal burn injury; omega 3 fatty acids; vitamin D; fish oil; chronic pain; chronic pain due to trauma
MeSH Terms: conditions — Burns; Chronic Pain | interventions — Fatty Acids, Omega-3; Fish Oils; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: 2x2 Factorial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- n-3 PUFA (O3FA) + Vitamin D3 (Experimental): 4g fish oil in 4 softgels (n-3 PUFA/O3FA) + 2000 IU Vitamin D3 in 1 capsule
  Interventions: Drug: Omega-3 fatty acids (fish oil); Drug: Vitamin D3 (cholecalciferol)
- n-3 PUFA (O3FA) Placebo + Vitamin D3 (Experimental): 4g of corn/soy oil blend in 4 softgels + 2000 IU Vitamin D3 in 1 capsule
  Interventions: Drug: Vitamin D3 (cholecalciferol); Drug: Omega-3 fatty acid placebo
- n-3 PUFAs (O3FA) + Vitamin D3 Placebo (Experimental): 4g fish oil in 4 softgels (n-3 PUFA/O3FA) + Vitamin D3 matching Placebo, an inert white powder placebo in 1 capsule
  Interventions: Drug: Omega-3 fatty acids (fish oil); Drug: Vitamin D3 (cholecalciferol) placebo
- n-3 PUFA (O3FA) Placebo + Vitamin D3 Placebo (Placebo Comparator): 4g n-3 PUFA/O3FA Matching Placebo, a corn/soy oil blend in 4 softgels + inert white powder Vitamin D3 matching placebo in 1 capsule
  Interventions: Drug: Vitamin D3 (cholecalciferol) placebo; Drug: Omega-3 fatty acid placebo

INTERVENTIONS:
Drug: Omega-3 fatty acids (fish oil) — 4 capsules comprising approximately 2 grams of Eicosapentaenoic acid/Docosahexaenoic acid (EPA/DHA) in a 3:2 ratio (this will require a total dose of 4 grams of fish oil). This will be administered daily, by mouth for 6 weeks
  Other Names: Fish oil; n-3 fatty acids
  Arms: n-3 PUFA (O3FA) + Vitamin D3; n-3 PUFAs (O3FA) + Vitamin D3 Placebo
Drug: Vitamin D3 (cholecalciferol) — 1 capsule containing 2000 IU of Vitamin D3. This will be administered daily, by mouth for 6 weeks following enrollment.
  Other Names: Cholecalciferol; Vitamin D3
  Arms: n-3 PUFA (O3FA) + Vitamin D3; n-3 PUFA (O3FA) Placebo + Vitamin D3
Drug: Vitamin D3 (cholecalciferol) placebo — 1 capsule containing inert substance. This will be administered daily, by mouth for 6 weeks following enrollment.
  Other Names: Placebo, inert white powder; Vitamin D3 Matching Placebo
  Arms: n-3 PUFA (O3FA) Placebo + Vitamin D3 Placebo; n-3 PUFAs (O3FA) + Vitamin D3 Placebo
Drug: Omega-3 fatty acid placebo — 4g of corn/soy oil blend in 4 softgels. This will be administered daily, by mouth for 6 weeks following enrollment.
  Other Names: Placebo, corn/soy oil soft gels; PUFA Matching Placebo
  Arms: n-3 PUFA (O3FA) Placebo + Vitamin D3; n-3 PUFA (O3FA) Placebo + Vitamin D3 Placebo

SUMMARY:
The goal of this study is to develop a safe, effective, and readily available treatment that will prevent chronic pain following Major Thermal Burn Injury (MThBI). Burn survivors are prone to develop chronic pain and there is an urgent unmet need for preventative treatments. The preventative treatments proposed for this study, Omega-3 Fatty Acids (O3FA) and Vitamin D have been selected given effectiveness across a range of painful musculoskeletal disorders and their wide availability and low cost. This study is a 2x2 factorial, double-blind, placebo-controlled randomized controlled trial test for the effectiveness of O3FA and Vitamin D to prevent chronic pain development. Burn survivors will be enrolled who have experienced thermal burns that cover less than 30% total body surface area that are severe enough to warrant surgical management, which represents the most common burn injury characteristics. Patients will be enrolled within 72 hours of their burn, and randomized via 1:1:1:1 allocation to receive placebo, O3FA, Vitamin D or both. The investigators will obtain blood samples on enrollment and at 6 weeks to assist in elucidating key mechanisms by which O3FA and Vitamin D reduce chronic pain following MThBI. Chronic pain severity, assessed with a 0-10 numeric rating scale at 6 weeks, 3 months, 6 months and 1 year will be entered into a repeated-measures model. Model estimated contrasts will serve as the primary outcome.

DETAILED DESCRIPTION:
Patients will be screened daily. Patients who meet eligibility criteria will be approached for participation. Patients interested in participating will proceed through informed consent. Once informed consent is obtained, an initial questionnaire will be administered, a blood draw will be performed to assess for baseline Vitamin D/O3FA concentration and immune profile. Then patients will be randomized into one of 4 treatment arms in 1:1:1:1 allocation. Patients will receive study drug for 6 weeks following burn injury. Adverse event monitoring will occur daily while inpatient and weekly once discharged from the hospital through 6 weeks. Patient compliance with the study drug will be assessed via patient-reported reported missing doses, pill counts at the end of the study, and a 6-week blood draw in which Vitamin D/O3FA levels and immune profile will be assessed. Patient-reported outcomes will be collected via follow-up survey at 6 weeks, 3 months, 6 months, and 1 year following burn injury.s, and 1 year following burn injury.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years and ≤ 65 years of age
* Admitted to burn center within 72 hours of thermal burn injury
* Estimated Total Body Surface area (TBSA) ≤ 30%
* Surgical team has plans for surgical management of the burn wound (e.g. xenograft and/or autograft).
* Patients experience a thermal burn injury, not an electrical or chemical burn.
* Has a telephone to receive follow-up calls.
* Able to speak and read English
* Resides within 150 miles of study site
* Alert and oriented
* Willing to take study medication for 6 weeks following enrollment
* Subjects are capable of giving informed consent.
* Predicted probability of chronic pain ≥ 0.3 when demographic parameters are entered into a logistic regression model developed from a previous cohort. (Initial pain score entered into this model will be based on the highest pain severity over the initial 24 hours of hospital admission).
* European American or African American

Exclusion Criteria:

* Unwilling to take study drug
* Allergy to fish oil or corn/soybean oil.
* Patient taking clopidogrel (Plavix)
* Patient taking warfarin or dabigatran.
* Substantial comorbid injury (e.g. long bone fracture)
* Pregnancy/Breastfeeding
* Prisoner status
* Chronic daily opioid use prior to burn (>20 mg oral daily morphine equivalents).
* Active psychosis, suicidal ideation, or homicidal ideation
* Requires an escharotomy or fasciotomy for the treatment of burn injury.
* Has a disorder of pain processing or diminished capacity to perceive pain (congenital insensitivity to pain)
* Known Child-Pugh liver disease severity classification B or C.
* Known chronic kidney disease stage 4 or higher (GFR≤29).
* Known Hemophilia A/B
* Known bleeding dyscrasia
* History of an inability to tolerate fish oil or corn/soybean oil.
* Severe gastroesophageal reflux disease
* No other history or condition that would, in the investigator's judgment, indicate that the patient would very likely be non-compliant with the study or unsuitable for the study (e.g. might interfere with the study, confound interpretation, or endanger patient).
* Intubated and sedated at time of enrollment.
* Hypersensitivity to Vitamin D3, ergocalciferol, calcitriol, alfacalcidol, calcipotriol
* Hypercalcemia (if not already completed, this will be assessed by clinical labs with albumin correction prior to enrollment).
* Hypervitaminosis
* Sarcoidosis
* Hyperphosphatemia
* Arteriosclerosis
* Active myocardial ischemia
* Frequent antacid use (calcium carbonate, cimetidine)
* Cholestyramine or Colestipol use
* Taking Vitamin D supplements in excess of 800 IU daily.
* Taking >1g of fish oil per day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Mauck, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University Of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared on request provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC) independently.
Time Frame: 12-36 months following publication
Access Criteria: Deidentified individual data that supports the results will be shared provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC independently.

RESULTS

PARTICIPANT FLOW:
Groups:
- n-3 PUFA (O3FA) + Vitamin D3: 4g fish oil in 4 softgels (n-3 PUFA/O3FA) + 2000 IU Vitamin D3 in 1 capsule
  Omega-3 fatty acids (fish oil): 4 capsules. This will be administered daily, by mouth for 6 weeks
  Vitamin D3 (cholecalciferol): 1 capsule containing 2000 IU of Vitamin D3. This will be administered daily, by mouth for 6 weeks following enrollment.
- n-3 PUFAs (O3FA) + Vitamin D3 Placebo: 4g fish oil in 4 softgels (n-3 PUFA/O3FA) + Vitamin D3 matching Placebo, an inert white powder placebo in 1 capsule
  Omega-3 fatty acids (fish oil): 4 capsules This will be administered daily, by mouth for 6 weeks
  Vitamin D3 (cholecalciferol) placebo: 1 capsule containing inert substance. This will be administered daily, by mouth for 6 weeks following enrollment.
Period: Overall Study
Arm/Group | n-3 PUFA (O3FA) + Vitamin D3 | n-3 PUFA (O3FA) Placebo + Vitamin D3 | n-3 PUFAs (O3FA) + Vitamin D3 Placebo | n-3 PUFA (O3FA) Placebo + Vitamin D3 Placebo
Started | 7 | 6 | 6 | 5
Completed | 5 | 4 | 4 | 3
Not Completed | 2 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- n-3 PUFA (O3FA) + Vitamin D3: 4g fish oil in 4 softgels (n-3 PUFA/O3FA) + 2000 IU Vitamin D3 in 1 capsule
  Omega-3 fatty acids (fish oil): 4 capsules This will be administered daily, by mouth for 6 weeks
  Vitamin D3 (cholecalciferol): 1 capsule containing 2000 IU of Vitamin D3. This will be administered daily, by mouth for 6 weeks following enrollment.
- Total: Total of all reporting groups
Arm/Group | n-3 PUFA (O3FA) + Vitamin D3 | n-3 PUFA (O3FA) Placebo + Vitamin D3 | n-3 PUFAs (O3FA) + Vitamin D3 Placebo | n-3 PUFA (O3FA) Placebo + Vitamin D3 Placebo | Total
Number analyzed (Participants) | 7 | 6 | 6 | 5 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (13.7) | 34.7 (12.6) | 26.9 (6.9) | 30.7 (9.39) | 32.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 1 | 5
  Male | 6 | 5 | 4 | 4 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black American | 3 | 4 | 3 | 3 | 13
  White American | 4 | 2 | 3 | 2 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 6 | 5 | 24
Education [Count of Participants; unit: Participants]
  Completed High School | 1 | 1 | 4 | 2 | 8
  Post-high school education | 3 | 4 | 1 | 2 | 10
  College Graduate or beyond | 3 | 1 | 1 | 1 | 6
Income [Count of Participants; unit: Participants]
  <$40,000/year | 1 | 1 | 3 | 2 | 7
  $40,000-$59,999/year | 1 | 2 | 0 | 1 | 4
  $60,000-$99,999/year | 0 | 1 | 0 | 1 | 2
  >$100,000/year | 2 | 0 | 0 | 0 | 2
  Refused/Don't know | 3 | 2 | 3 | 1 | 9
Total Body Surface Area Burned [Mean (Standard Deviation); unit: Percent total body surface area burned] — Total body surface area affected by the burn
  Percent total body surface area burned | 4.8 (4.01) | 7.9 (6.4) | 6.0 (4.7) | 5.3 (3.9) | 6.1 (4.7)
Type of Thermal Burn [Count of Participants; unit: Participants]
  Flame | 4 | 3 | 2 | 3 | 12
  Contact | 0 | 0 | 1 | 0 | 1
  Scald | 0 | 2 | 2 | 2 | 6
  Other | 2 | 1 | 1 | 0 | 4
  Not reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Review of Treatment-Related Adverse Events
Description: A primary objective of this pilot study is to ensure safety of both treatments as well as combined. A qualitative review of treatment-related adverse events will be performed and a determination about the degree of relatedness of each adverse event with the intervention using CTCAE criteria will be made as CTCAE criteria assesses relatedness to therapy. Investigator reviewing the details of each adverse event rated the likelihood of relatedness to the study drug on a scale: (unrelated, unlikely, possible, probably, definitely).
Time Frame: 6 weeks following burn injury
Population: Enrolled participants who initiated study treatment
Measure: Number; unit: adverse events
Groups:
- n-3 PUFA (O3FA) + Vitamin D3: 4g fish oil in 4 softgels (n-3 PUFA/O3FA) + 2000 IU Vitamin D3 in 1 capsule
  Omega-3 fatty acids (fish oil): 4 capsules.This will be administered daily, by mouth for 6 weeks
  Vitamin D3 (cholecalciferol): 1 capsule containing 2000 IU of Vitamin D3. This will be administered daily, by mouth for 6 weeks following enrollment.
- n-3 PUFAs (O3FA) + Vitamin D3 Placebo: 4g fish oil in 4 softgels (n-3 PUFA/O3FA) + Vitamin D3 matching Placebo, an inert white powder placebo in 1 capsule
  Omega-3 fatty acids (fish oil): 4 capsules. This will be administered daily, by mouth for 6 weeks
  Vitamin D3 (cholecalciferol) placebo: 1 capsule containing inert substance. This will be administered daily, by mouth for 6 weeks following enrollment.
Arm/Group | n-3 PUFA (O3FA) + Vitamin D3 | n-3 PUFAs (O3FA) + Vitamin D3 Placebo | n-3 PUFA (O3FA) Placebo + Vitamin D3 | n-3 PUFA (O3FA) Placebo + Vitamin D3 Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
adverse events
  Unrelated | 3 | 4 | 2 | 2
  Unlikely Related | 1 | 3 | 2 | 3
  Possibly Related | 1 | 2 | 0 | 0
  Probably Related | 0 | 0 | 0 | 0
  Definitely Related | 1 | 1 | 0 | 0

2. Primary Outcome: Percent of Participants Who Are Compliant With Follow-up (Feasibility)
Description: The primary objective of this pilot study is to ensure that the investigators are able to make follow-up assessments on a majority of participants. The percent of participants who are compliant with follow-up will be determined 6 weeks following major thermal burn injury. Feasibility is defined as >80% of enrolled participants at 6 weeks following Major Thermal Burn Injury (MThBI).
Time Frame: 6 weeks following burn injury
Population: After informed consent, initial survey completion, and randomization, 2 participants in the n-3 PUFA (O3FA) + Vitamin D3 dropped out of the study and were not included in these analyses.
Measure: Number; unit: percentage of participants
Groups:
- n-3 PUFAs (O3FA) + Vitamin D3 Placebo: 4g fish oil in 4 softgels (n-3 PUFA/O3FA) + Vitamin D3 matching Placebo, an inert white powder placebo in 1 capsule
  Omega-3 fatty acids (fish oil): 4 capsules.This will be administered daily, by mouth for 6 weeks
  Vitamin D3 (cholecalciferol) placebo: 1 capsule containing inert substance. This will be administered daily, by mouth for 6 weeks following enrollment.
Arm/Group | n-3 PUFA (O3FA) + Vitamin D3 | n-3 PUFA (O3FA) Placebo + Vitamin D3 | n-3 PUFAs (O3FA) + Vitamin D3 Placebo | n-3 PUFA (O3FA) Placebo + Vitamin D3 Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 5
percentage of participants | 100 | 50 | 83.3 | 80

3. Primary Outcome: By Group Efficacy Estimates Over Year Following Thermal Burn Injury
Description: Estimates of efficacy will be obtained via repeated measures analysis of pain severity over the 1 year following injury using mixed effects models. Pain will be assessed using a 0-10 numeric rating scale with 0 indicating no pain and 10 indicating pain as severe as you can imagine. Higher scores represent worse outcome. These values (collected in identical fashion over 1 year following burn injury) will be entered into a linear mixed model, and overall effect estimates (beta coefficients) among groups will be determined. Final model was a piece-wise linear mixed model, with a cut-point at 6 weeks. Mixed models were adjusted for age, sex, race, initial pain severity. Every 1 unit change in beta coefficient represents a 1 unit change in pain severity on the 0-10 numeric rating scale.
Time Frame: Over 1 year following MThBI
Population: Given the 2x2 factorial design, comparisons were made to assess the differences between one treatment and placebo regardless of the other treatment. E.g. groups were combined to assess whether there was any difference between Vitamin D and placebo regardless of O3FA treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Omega-3: Omega 3 active treatment
- No Omega 3 Treatment: Omega 3 placebo
- Vitamin D: Vitamin D active treatment
- No Vitamin D Treatment: Vitamin D placebo
Arm/Group | Omega-3 | No Omega 3 Treatment | Vitamin D | No Vitamin D Treatment
Number analyzed (Participants) | 13 | 11 | 13 | 11
score on a scale
  Baseline (Day 1) | 7.19 (1.15) | 7.57 (1.83) | 7.01 (1.72) | 7.65 (1.14)
  Week 1: number analyzed (Participants) | 13 | 10 | 12 | 11
  Week 1 | 5.7 (2.21) | 5.50 (2.21) | 5 (2.65) | 6.09 (2.21)
  Week 2: number analyzed (Participants) | 11 | 10 | 10 | 11
  Week 2 | 4.5 (2.99) | 3.8 (3.01) | 3.22 (2.33) | 4.91 (3.27)
  Week 3: number analyzed (Participants) | 11 | 10 | 11 | 10
  Week 3 | 2.0 (2.45) | 2.8 (2.49) | 1.9 (1.97) | 2.90 (2.85)
  Week 4: number analyzed (Participants) | 11 | 9 | 10 | 10
  Week 4 | 1.73 (2.20) | 2.33 (1.94) | 1.6 (1.78) | 2.4 (2.32)
  Week 5: number analyzed (Participants) | 11 | 7 | 8 | 10
  Week 5 | 1.22 (1.48) | 1.43 (1.27) | 1 (1.15) | 1.56 (1.51)
  Week 6: number analyzed (Participants) | 10 | 8 | 9 | 9
  Week 6 | 1.6 (1.58) | 1.57 (2.94) | 0.75 (1.04) | 2.33 (2.65)
  Month 3: number analyzed (Participants) | 7 | 5 | 7 | 5
  Month 3 | 0.67 (1.15) | 0.33 (0.58) | 0.25 (0.5) | 1.0 (1.41)
  Month 6: number analyzed (Participants) | 7 | 6 | 6 | 7
  Month 6 | 1.14 (1.46) | 0.33 (0.82) | 0.67 (1.03) | 0.86 (1.46)
  Month 12: number analyzed (Participants) | 5 | 4 | 5 | 4
  Month 12 | 1.2 (2.17) | 0.5 (1.0) | 0.6 (0.89) | 1.25 (2.5)
Statistical Analysis 1: Comparison: Vitamin D vs No Vitamin D Treatment; Test type: Superiority; p = 0.276, Mixed Models Analysis — The final, adjusted p-value threshold of 0.0492, using the O'Brien-Fleming approach, allows for a statistical "penalty" to be assessed because of the interim analysis; The model was adjusted for age, sex, race, treatment interaction, initial pain severity, and total body surface area burned; Slope = -0.84, 95% CI 2-sided [-2.32 to 0.63]
Statistical Analysis 2: Comparison: Omega-3 vs No Omega 3 Treatment; Test type: Superiority; p = 0.336, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Slope = 0.72, 95% CI 2-sided [-0.71 to 2.14]
Statistical Analysis 3: Comparison: Vitamin D vs No Vitamin D Treatment; Sensitivity analysis adjusting for an influential observation (using the dfbeta approach) that could produce spurious results from a small trial dataset; Test type: Superiority; p = 0.004, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Slope = -2.33, 95% CI 2-sided [-3.76 to -0.9]
Statistical Analysis 4: Comparison: Omega-3 vs No Omega 3 Treatment; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.139, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Slope = 0.92, 95% CI 2-sided [-0.25 to 2.09]

4. Secondary Outcome: Sex Differences in Treatment Response Based on Pain Scores
Description: Examines existence of gender-based treatment response differences in pain severity measured by a 0-10 numeric rating scale where 0 is no pain and 10 is the most severe pain. Higher scores reflect greater pain (poor outcome).
Time Frame: 6 weeks following burn injury
Population: The population included were participants who responded to the graft site pain severity question at the 6-week follow-up surveys. Treatment assignment of Omega-3 fatty acids or no Omega-3 fatty acids was considered independent of Vitamin D treatment. Treatment assignment of Vitamin D or no Vitamin D treatment was considered independent of Omega-3 fatty acid treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega-3 | No Omega 3 Treatment | Vitamin D | No Vitamin D Treatment
Number analyzed (Participants) | 10 | 7 | 8 | 9
units on a scale
  Male: number analyzed (Participants) | 7 | 5 | 6 | 6
  Male | 1.43 (1.81) | 1.80 (3.49) | 0.33 (0.81) | 2.83 (3.01)
  Female: number analyzed (Participants) | 3 | 2 | 2 | 3
  Female | 2.00 (1.00) | 1.00 (1.42) | 2 (0) | 1.33 (1.52)

5. Secondary Outcome: General Mental Health as Measured by the Short Form (SF)-12 General Mental Health Component Scores
Description: Assessment of mental health will be determined by the short form (SF)-12 mental component score. The short form SF-12 Health Survey is a 12-item participant completed questionnaire to measure general health. It includes a mental component score (MCS): ranging from 0 to 100 points. Low values represent a poor health state and high values represent a good mental health.
Time Frame: 6 weeks following burn injury
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 | No Omega 3 Treatment | Vitamin D | No Vitamin D Treatment
Number analyzed (Participants) | 10 | 7 | 8 | 9
score on a scale | 49.98 (9.98) | 48.29 (10.79) | 52.80 (6.37) | 46.16 (11.92)

6. Secondary Outcome: General Physical Health by Treatment Group Measured by the SF-12 General Physical Health Component Scores
Description: Assessment of physical health will be determined by the SF-12 physical component score. The SF-12 Health Survey is a 12 item participant completed questionnaire to measure general health. It includes a physical component score (PCS): ranging from 0 to 100 points. Low values represent a poor physical health and high values represent a good physical health.
Time Frame: 6 weeks following burn injury
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 | No Omega 3 Treatment | Vitamin D | No Vitamin D Treatment
Number analyzed (Participants) | 10 | 7 | 8 | 9
score on a scale | 40.84 (6.25) | 40.12 (6.40) | 40.83 (3.85) | 40.29 (7.86)

7. Secondary Outcome: Pain Interference by Treatment Group Measured by the Brief Pain Inventory
Description: The degree to which pain interferes with important life function will be determined by the Brief Pain Inventory. This is a validated, self-reported scale that measures the severity of pain based on the average pain experienced and assesses impact of pain across 7 domains of life function (e.g., enjoyment of life, relationships, normal work). The total severity scores range from 0 (no interference) to 70 (maximum interference). Higher scores reflect greater pain interference.
Time Frame: 6 weeks following burn injury
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 | No Omega 3 Treatment | Vitamin D | No Vitamin D Treatment
Number analyzed (Participants) | 10 | 7 | 8 | 9
score on a scale | 11.60 (12.76) | 13.71 (20.30) | 5.5 (6.85) | 18.67 (19.03)

ADVERSE EVENTS:
Time Frame: After randomization through 6 weeks of active treatment
Description: Participants responded via weekly surveys to assess adverse events
Arm/Group | n-3 PUFA (O3FA) + Vitamin D3 | n-3 PUFA (O3FA) Placebo + Vitamin D3 | n-3 PUFAs (O3FA) + Vitamin D3 Placebo | n-3 PUFA (O3FA) Placebo + Vitamin D3 Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 3/7 | 1/6 | 3/6 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | n-3 PUFA (O3FA) + Vitamin D3 (N=7) | n-3 PUFA (O3FA) Placebo + Vitamin D3 (N=6) | n-3 PUFAs (O3FA) + Vitamin D3 Placebo (N=6) | n-3 PUFA (O3FA) Placebo + Vitamin D3 Placebo (N=5)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Mild reduction in hemoglobin concentration
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Medication administration error (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Medication administration/dosing error
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood Swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated PTT (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral Sore (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination because of pandemic delays

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT03313076/Prot_SAP_000.pdf